CLINICAL TRIAL: NCT00802698
Title: The Effect of Transcorneal Stimulation in Cases of Central Retinal Artery Occlusion Using a New Waveform
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-039
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Central Retinal Artery Occlusion
Keywords: Biphasic waveform; Central retinal artery occlusion; To describe the effect of Transcorneal Electrical Stimulation (TES) with a non conventional biphasic bipolar waveform; in central retinal artery occlusion
MeSH Terms: conditions — Retinal Artery Occlusion

ARMS (1):
- Group 1 (Experimental)
  Interventions: Device: Transcorneal electric stimulation; Device: Transcorneal stimulation

INTERVENTIONS:
Device: Transcorneal electric stimulation — central artery occlusion
  Other Names: TES
Device: Transcorneal stimulation — new waveform
  Other Names: TES
Device: transcorneal electric stimulation — Novel waveform central artery occlusion
  Other Names: TES

SUMMARY:
The purpose of this study is to describe the effect of transcorneal electrical stimulation (TES) with a non conventional biphasic bipolar waveform in central retinal artery occlusion

DETAILED DESCRIPTION:
Patients with acute central retinal artery occlusion (CRAO) generally present with a history of painless visual loss that occurred over several seconds. In some instances amaurosis fugax is also present. At the time of initial examination, visual acuity in 90% of patients with CRAO can vary from counting fingers to light perception. Acute CRAO is considered an emergency situation, and therapy must be started as soon as possible. There are different reports where different treatments were proved for the acute phase for example: ocular massage, anterior chamber paracentesis, intravenous mannitol, acetazolamide, hyperbaric oxygenation, microcatheter urokinase infusion, and carbogen 1,2,3. Electrophysiological occlusion of the ophthalmic artery, central retinal artery occlusion, or central retinal vein has a profound impact on the ERG. ERG can provide an objective assessment of severity if occlusion occurs, the b wave is eliminated and a reduction in the "a" wave can be observed.

In addition, a traumatic optic neuropathy, together with retinal ganglion cell death, can induce a loss of vision which progresses rapidly within several hours l. It is known that the visual prognosis following treatment of acute central retinal artery occlusion is not as good as we would like 2; the patient must go to any emergency department to be treated immediately3, in order to preserve maximal visual function. It has been prove that the retinal function recovers after an ischemic event lasting up to 97 minutes, 4 and irreparable damage may occur after 105 minutes. This is why this study intervene during the chronic phase between 4 hrs and 14 days; where demonstrable clinical improvements in the magnitude of retinal damage where seen5, 6, 7 However recently research reports have shown that, electrical stimulation can rescue injured retinal ganglion cells from death cells and can preserve visual function after an optic nerve crush. 8 There is no ideal treatment in the chronic phase of the CRAO. That is the reason why most recent papers suggest different treatment approaches in the chronic phase of this pathology. One of these treatments that were described is the application of electrical stimulation on the patient's cornea who present with CRAO. It has been reported in the literature that transcorneal, retinal 9,10 or cerebral visual cortex 11 electrical stimulation (ES) results in evoked visual sensations (phosphenes),6,9,10,12 however, this intervention requires surgical electrode implantation.

ELIGIBILITY:
Inclusion Criteria:

* central retinal Artery occlusion
* no retinal diseases associated
* visual acuity in other eye better than 20/200

Exclusion Criteria:

* Branch retinal artery occlusion

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Baseline, Final

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Jessica Lopez-Miranda, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- APEC, México, Mexico